CLINICAL TRIAL: NCT01524211
Title: Evaluation of Branch Endografts in the Treatment of Aortic Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: William Cook Australia (Industry); Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE G110081
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Thoracoabdominal Aortic Aneurysm; Aortic Arch Aneurysm
Keywords: Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aneurysm, Aortic Arch; Aortic Aneurysm

STUDY DESIGN:
Intervention Model Description: Zenith t-Branch Subject Cohort: All eligible subjects will receive treatment with the investigational t-Branch Endovascular Graft. (Total 225 subjects)
  Terumo Arch Branch Cohort: All eligible subjects will receive treatment with the investigational Terumo Arch Branch Endovascular Graft. (Total 10 Subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Single Treatment Arm-Zenith t-Branch Cohort (Experimental): Zenith t-Branch Cohort:Those subjects eligible for enrollment will receive endovascular treatment with the investigational Zenith t-Branch Endovascular Graft.
  Interventions: Device: Zenith® t-Branch
- Single Treatment Arm-Terumo Arch Branch Cohort (Experimental): Terumo Arch Branch Cohort:Those subjects eligible for enrollment will receive endovascular treatment with the investigational Terumo Arch Branch Endovascular Graft.
  Interventions: Device: Terumo Arch Branch

INTERVENTIONS:
Device: Zenith® t-Branch — The t-Branch Endovascular Graft (Zenith® t-Branch) is a tubular graft with four branches and a covered stent at the proximal end that contains barbs for additional fixation of the device. The purpose of the branches is to allow uninterrupted blood flow to visceral vessels of the aorta. The graft is designed to be connected with celiac, superior mesenteric and two renal arteries via self-expanding covered bridging stents. Although the standard Zenith t-Branch has four branches, it is anticipated that a small number of custom-made three branch devices will be included in this study for those patients in whom one of the visceral vessels is chronically thrombosed.
  Arms: Single Treatment Arm-Zenith t-Branch Cohort
Device: Terumo Arch Branch — The Arch Branch endograft is a custom-made endograft based on the Relay thoracic stent graft platform. The device is intended to land proximally in the ascending aorta just distal to the sinotubular junction, and distally either in the native thoracic aorta for focal arch pathologies, or more extensive pathologies either extended with another commercially available thoracic endograft or mated to a pre-existing thoracic endograft, which would serve as a distal landing zone. It is constructed of polyester graft material (same as those used for the Terumo Relay Plus or Pro) sewn to self-expanding nitinol stents with suture. The graft is fully stented to provide stability and the expansile force necessary to open the lumen of the graft during deployment. Additionally, the stents provide the necessary attachment and seal of the graft to the aortic wall.
  Arms: Single Treatment Arm-Terumo Arch Branch Cohort

SUMMARY:
Zenith t-Branch Study Cohort: The purpose of this study is to collect information on the Cook Zenith t-Branch endovascular stent-graft system and the Terumo Arch Branch for the treatment of aortic aneurysms.

Terumo Arch Branch Study Cohort: The purpose of this additional study arm to the current IDE clinical trial is to collect a priori information on the Terumo Arch Branch Endograft for the treatment of proximal thoracic aortic pathologies that cannot be treated with conventional thoracic endografts.

DETAILED DESCRIPTION:
Study Update as of 3/31/2025; 186 subjects successfully have been implanted with the Zenith t-Branch Device and 1 subject has been implanted with the Arch Branch to date and recruitment is ongoing.

ELIGIBILITY:
Zenith t-Branch Eligibility Criteria:

Inclusion Criteria

The patient must have one of the following:

1. Degenerative, atherosclerotic thoracoabdominal, suprarenal and juxtarenal aortic aneurysms (fusiform or saccular):≥55mm in diameter in a male or ≥50mm in diameter in a female, or
2. Thoracoabdominal aortic aneurysm with a history of growth ≥0.5 cm per year, or
3. Penetrating ulcers: ≥20mm in depth or
4. Chronic type B aortic dissections: ≥50mm total aortic diameter or
5. Symptomatic pathology (aneurysm, ulcer or chronic dissection) of any size.

Additional criteria for LP material

• Iliofemoral access vessels <8mm or with significant atherosclerotic occlusive disease that would require an iliac conduit as determined by the Principle Investigator

Exclusion Criteria

General Criteria

1. Life-expectancy less than 12 months
2. Refusal to receive blood products
3. Age <18 years
4. Pregnant or breastfeeding or planning on becoming pregnant within 60 months
5. Unwilling to comply with the follow-up schedule
6. Inability or refusal to give informed consent by subject and/or Legally Authorized Representative (LAR); should one be utilized

Medical Criteria

1. Uncontrolled systemic infection
2. Untreatable malignancy
3. Uncontrollable anaphylaxis to iodinated contrast
4. Known allergy(ies) to device materials

Anatomic Criteria

1. Any pathology of mycotic origin
2. Aortic fistulous communication with non-vascular structure (e.g. esophagus, bronchial)
3. Inability to insert the Zenith® t-Branch device through iliofemoral approach
4. Proximal and distal neck angle less than 90 degrees relative to the long axis of the aneurysm
5. Proximal landing zone length <25mm to allow secure fixation and seal
6. Proximal landing zone diameter of <24mm or >42mm
7. Distal landing zone length <25mm in the abdominal aorta or <20mm in the iliac arteries
8. Distal landing zone diameter of <14mm or >30mm in the abdominal aorta, or <7mm or >28mm in the iliac arteries

Terumo Arch Branch Eligibility Criteria

Inclusion Criteria

The subject must have one of the following:

1. Degenerative, atherosclerotic aneurysm involving the ascending aorta, aortic arch or proximal descending aorta ≥55 mm in diameter or > 50 mm with a history of growth ≥5 mm in the last 6 months, or
2. Penetrating ulcers: ≥20 mm in depth, or
3. Chronic aortic dissections: ≥50mm total aortic diameter. AND Prohibitive or high-risk for standard open surgical repair, defined as having one or more of the following pre-existing conditions.

   1. Age >85 years old.
   2. Prior median sternotomy (for any reason).
   3. Prior open or endovascular thoracic aortic repair.
   4. Severe aortic calcification.
   5. Severe occlusive disease of one or more arch vessels.
   6. Moderate-severe COPD (FEV1 <80% predicted).
   7. Severe CKD (Stage 3 or greater, eGFR <60 mL/min).
   8. LV dysfunction.
   9. Chronic steroid or immunosuppressive use.
   10. History of increased risk of bleeding.
   11. Neurocognitive deficits that may significantly impact postoperative rehabilitation.
   12. Musculoskeletal conditions that may significantly impact postoperative rehabilitation.

Exclusion Criteria

General Criteria

1. Life expectancy <1 year.
2. Refusal to receive blood products.
3. Age <18 years.
4. Pregnant, breastfeeding, or planning to become pregnant within 60 months.
5. Unwilling to comply with the follow-up schedule.
6. Inability or refusal to give informed consent by subject and/or Legally Authorized Representative (LAR); should one be utilized.
7. Willingness to travel, if needed, to participate in a manufacturer-sponsored clinical trial at another institution.

Medical Criteria

1. Pending cardiac surgery.
2. Untreatable severe, symptomatic coronary or valvular disease.
3. Prior mechanical aortic valve replacement (not bioprosthetic).
4. History of TAVR (Transcatheter Aortic Valve Replacement)
5. Severe, calcific aortic valvular stenosis.
6. Uncontrolled systemic infection.
7. Untreatable malignancy with <1 year expected survival.
8. Uncontrollable anaphylaxis to iodinated contrast.
9. Known allergy(ies) to device materials. (i.e. polyester, nitinol).

Anatomic Criteria

1. Any pathology of mycotic origin.
2. Aortic fistulous communication with non-vascular structure (e.g. esophagus, bronchial).
3. Acute (<2 weeks) aortic dissection.
4. Type A dissection.
5. Symptomatic or ruptured pathology.
6. Anatomy suitable for repair using commercially-available endograft.
7. Inability to insert the Arch Branch endograft through an iliofemoral approach.
8. Untreated, known extracranial carotid stenosis >80%.
9. Ascending aortic angulation with radius of curvature <15mm in the intended landing zone.
10. Proximal aortic landing zone length <25 mm.
11. Proximal aortic landing zone diameter of >43mm or <28 mm.
12. Distal aortic landing zone diameter <20 mm.
13. Total length along the outer curve from the distal coronary to the proximal edge of the brachiocephalic trunk <70mm.
14. Target arch vessels:
15. Distal branch landing zone dimensions: I. Brachiocephalic trunk (innominate artery, BCT): Diameter >24 mm or <6 mm, length <15 mm. ii. Common carotid artery: Diameter <6 mm, length <25mm. iii. Subclavian artery: Diameter <6 mm, length <25mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2012-01-25 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Early Mortality & Stroke | 30 days post implant of the branch endografts
  The primary aim of this study is to determine the rate of early mortality and stroke after branch endograft treatment.

SECONDARY OUTCOMES:
Rates of Neurologic Complications/Late Branch Vessel Patency | Day 0-Day 30 (Early) Day 31-1825 (Late)
  The secondary aims of this study are to determine the rates of neurologic complications and late branch/target vessel patency, type I and III endoleaks and secondary interventions after branch endograft treatment. In those subjects enrolled in the t-Branch cohort we will evaluate the fractional/proportional/percent applicability/eligibility of the (standard, off-the-shelf) Zenith® t-Branch in all patients who present with thoracoabdominal aortic aneurysms.

CONTACTS AND LOCATIONS:
Overall Officials: W. Anthony Lee, MD, Principal Investigator — Lynn Heart and Vascular Institute, Boca Raton Regional Hospital
Locations (1):
- Baptist Health South Florida|Boca Raton Regional Hospital (BRRH), Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702